CLINICAL TRIAL: NCT06057935
Title: ICARuS II (Intraperitoneal Chemotherapy After cytoReductive Surgery): A Multicenter, Randomized Phase II Trial of Normothermic Intraperitoneal Chemotherapy and Intravenous Chemotherapy After Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy for Malignant Peritoneal Mesothelioma
Brief Title: A Study of Additional Chemotherapy After Surgery for People With Malignant Peritoneal Mesothelioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-145
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Malignant Peritoneal Mesothelioma; Peritoneal Mesothelioma; Mesothelioma; Mesothelioma, Malignant; Malignant Mesothelioma
Keywords: Malignant Peritoneal Mesothelioma; Peritoneal Mesothelioma; Mesothelioma; Mesothelioma, Malignant; Malignant Mesothelioma; ICARuS II; Memorial Sloan Kettering Cancer Center; 23-145
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IVC arm (Experimental): Pemetrexed and cisplatin will be administered intravenously for a total of 4 to 6 cycles. Participants will receive 4 cycles, but can receive up to 6 cycles based on clinician discretion. Substitution with carboplatin allowed for pre-existing impairment of hearing, renal function, or neuropathy.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- NIPC arm (Active Comparator): After completion of hyperthermic intraperitoneal chemotherapy/HIPEC, an intraperitoneal catheter with a subcutaneous reservoir will be inserted through the abdominal wall. When the participant's condition is considered stable by the physicians, the NIPC will be started. Pemetrexed and either cisplatin or carboplatin will be administered through the intraperitoneal port.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed will be administered intravenously
Drug: Cisplatin — Cisplatin will be administered intravenously
Drug: Carboplatin — Possible substitution with carboplatin based on clinician discretion

SUMMARY:
The purpose of this study is to find out whether intraperitoneal or intravenous chemotherapy given after cytoreductive surgery and HIPEC are effective treatments for people with malignant peritoneal mesothelioma. Outcomes will be compared by observing intraperitoneal versus intravenous treatments to analyze if one is better than the other.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years or older, both sexes.
* Clinical diagnosis of MPM at enrolling institution.
* Prior to randomization, intraoperative pathologic confirmation of epithelioid MPM at enrolling institution.
* Complete or near-complete CRS achieved.
* Patient must be planning to undergo complete cytoreduction of all peritoneal disease.
* ECOG performance status ≤ 1.
* Hematology: ANC ≥ 1,500/µl.
* Platelets > 75,000/µl.
* Adequate renal function: creatinine < 1.5× the upper limit of normal (ULN) or calculated creatinine clearance of ≥50 ml/min.
* Adequate hepatic function: bilirubin < 1.5 mg/dl (except in patients with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL).
* Women of childbearing potential with a negative pregnancy test result (urine or blood) who agree to use an effective contraceptive method. Reliable contraception should be used from trial screening and must be continued throughout the study. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant.
* A man participating in this study must agree to utilize a reliable barrier form of contraception for the duration of the study
* Signed and dated written informed consent to participate in this clinical trial must be obtained prior to any study procedure.

Exclusion Criteria:

* Subjects who have previously undergone intraperitoneal chemotherapy or systemic chemotherapy for peritoneal mesothelioma.
* Subjects who have previously received platinum-containing chemotherapy regimens.
* Subjects with preoperative or intraoperative biopsy consistent with sarcomatoid mesothelioma, well-differentiated papillary mesothelioma, or benign multicystic mesothelioma.
* Other prior malignancies, except for cured non-melanoma skin cancer, curatively treated in situ carcinoma of the cervix, adequately treated malignancies for which there has been no evidence of activity for more than three years, or indolent tumors for which observation over two years is a reasonable option.
* High suspicion for extra-abdominal metastases.
* Women who are pregnant or lactating.
* Active coronary artery disease (defined as unstable angina or a positive cardiac stress test). Subjects with a history of coronary artery disease may be included if they have had a normal stress test within 60 days of enrollment or are determined by a cardiologist to be of acceptable perioperative risk.
* Uncontrolled hypertension defined as >140/90 and not cleared for surgery at the time of consent.
* New York Heart Association (NYHA) Class II or higher congestive heart failure; restrictive or obstructive pulmonary disease that would limit study compliance or place the patient at unacceptable risk for participation in the study.
* History of cerebrovascular disease that would limit study compliance or place the patient at unacceptable risk for participation in the study.
* Subjects with other concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study or place them at an unacceptable risk for participation in the study.
* Patients with known cisplatin, carboplatin, pemetrexed or mitomycin allergy.
* Evidence of extensive intraperitoneal adhesions at the time of surgery which prohibits intraperitoneal therapy, as determined by the operating surgeon.
* Any condition that would preclude the ability to deliver appropriate IP therapy.
* Use of an oral medication, lacking a suitable non-oral substitute, that if held for up to ten days, would be felt an unacceptable risk by the investigator.
* Life expectancy < 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2028-09-21 (Estimated); Study Completion 2028-09-21 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to 24 months
  Progression Free Survival in the two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Garrett Nash, MD, Principal Investigator — Memorial Sloan Kettering Cancer
Locations (13):
- United States (13):
  - University of Chicago (Data Collection Only), Chicago, Illinois
  - University of Michigan (Data Collection Only), Ann Arbor, Michigan
  - Washington University (Data Collection Only), St Louis, Missouri
  - University of Nebraska (Data collection only), Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Rutgers University (Data Collection Only), New Brunswick, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activites), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Allegheny Health Network (Data Collection Only), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org